CLINICAL TRIAL: NCT07127406
Title: The Frequency of Euglycemic Diabetic Ketoacidosis in Patients Using Sodium- Glucose Cotransporter-2 (SGLT-2) Inhibitor Admitted to the Postoperative Care Unit and Its Effect on Postoperative Outcomes: A Prospective Observational Study
Brief Title: Postoperative Euglycemic Ketoacidosis Frequency in Sodium-Glucose Cotransporter-2 Inhibitor Users
Acronym: SGLT-2I
Status: Active, not recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Zeynep Turan Civraz, Assoc.Prof., Kocaeli City Hospital
Other Study IDs: KSH-01
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Ketoacidosis; Postoperative Care
Keywords: euglycemic diabetic ketoacidosis; SGLT-2 Inhibitors
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Euglycemic Diabetic ketoacidosis: Patients who develops euglycemic diabetic ketoacidosis during postoperative follow up will be included this group
- No euglycemic diabetic ketoacidosis: Patients who do not develop euglycemic diabetic ketoacidosis during postoperative follow up

SUMMARY:
The goal of this observational study is to determine the frequency of postoperative euglycemic diabetic ketoacidosis (EDKA) in patients receiving Sodium- Glucose Cotransporter-2 (SGLT-2) inhibitors. The main questions it aims to answer are:Is the use of SGLT-2 inhibitors a factor that increases the incidence of euglycemic diabetic ketoacidosis in patients in the perioperative period or what conditions in the perioperative period cause EDKA in patients on SGLT-2 inhibitors?

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is one of the leading diseases with serious social and economic consequences and high mortality and morbidity. Diabetic ketoacidosis is a serious complication of DM. Diabetic ketoacidosis (DKΑ) is typically associated with type 1 diabetes. It also occurs in type 2 diabetes under conditions of extreme stress, such as severe infection, trauma, cardiovascular or other emergencies, in association with the use of SGLT2 inhibitors, or as a manifestation of type 2 diabetes in some populations, a disorder called ketosis-prone diabetes mellitus. Treatment of DKA is a clinical emergency. Hyperglycemia (blood glucose >250 mg/dL), metabolic acidosis (pH<7.3), ketosis (ketonemia or ketonuria) are the diagnostic criteria for diabetic ketoacidosis . Although elevated glucose is considered to be the sine qua non of diabetic ketoacidosis, diabetic ketoacidosis may be observed in a group of patients with blood glucose <250 mg/dL. This condition is called euglycemic diabetic ketoacidosis (EDKA). Although it is a rare condition, a normal glucose level may lead to delayed treatment and consequently increased morbidity and mortality, as it may distract from the diagnosis. The pathophysiology of this clinical condition is unclear and has been reported in patients with type 1 and type 2 diabetes with SGLT2 inhibitor use.Factors that increase the risk of EDKA in patients using SGLT2 inhibitors include vomiting, dehydration, infection, surgery, low-carbohydrate diet, and underlying malignancy, which are common conditions in surgical patients. In recent years, with the increase in the frequency of EDKA in the perioperative period, it is recommended by the US Food and Drug Administration to discontinue this group of drugs at least 3-4 days before surgery.

The use of SGLT2 inhibitors is rapidly increasing in patients diagnosed with diabetes, heart failure and chronic kidney disease due to their nephroprotective and cardioprotective effects. SGLT-2 inhibitor use is also more common in the surgical patient population. The number of patients operated in the operating rooms of our hospital in 2023 is 23502. The number of patients admitted to the postoperative care unit (PACU) since the opening of our hospital is 3135. The majority of these patients have hypertension, diabetes mellitus, chronic heart failure and other comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* patients who is 18 years old and older
* Patients using SGLT-2 inhibitors and admitted to the postoperative intensive care unit after surgery.

Exclusion Criteria:

* Patients who is younger than 18 years old
* Patients who undergoes emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the postoperative intensive care unit will be evaluated for inclusion in the study. patients over the age of 18 years who use SGLT-2 inhibitors in the preoperative period will be included in the study. they will be followed up for the development of euglycemic diabetic ketoacidosis after informed consent is obtained from them or their families.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of diabetic ketoacidosis in Postoperative care unit among patients who receives SGLT-2 inhibitor | 24 hours after surgery
  Patients receiving SGLT-2 inhibitors will be follow up in postoperative care unit.

SECONDARY OUTCOMES:
Length of ICU stay | 30 day
  Length of ICU stay will be recorded.
Length of hospital stay | 30 days
  Length of hospital stay will be recorded
ICU readmission | 30 days
  ICU readmission will be recorded
30 day mortality | 30 days
  Mortality will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Z Turan Cıvraz, Assoc. Prof., Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided